CLINICAL TRIAL: NCT04057586
Title: Postoperative Cognitive Dysfunction After Intubated and Non-intubated Thoracic Surgery: a Randomized Controlled Trial
Brief Title: Cognitive Recovery Between Intubated and Non-intubated Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201904071RINC
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2019-06

CONDITIONS: Cognition
Keywords: postoperative cognition; nonintubated thoracic surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonintubated (Experimental): Nonintubated thoracoscopic surgery
  Interventions: Procedure: Nonintubated
- Intubated (Active Comparator): Intubated thoracoscopic surgery
  Interventions: Procedure: Intubated

INTERVENTIONS:
Procedure: Nonintubated — During surgery, patient is deeply sedated and respiration is maintained by spontaneous breath under the nasal high flow oxygen support.
  Arms: Nonintubated
Procedure: Intubated — During surgery, patient received standard general anesthesia and respiration is maintained by using mechanical ventilation.
  Arms: Intubated

SUMMARY:
In this randomized controlled trial, we aim to investigate whether the avoidance of mechanical ventilation by application of nonintubated thoracoscopic surgery improves intraoperative cerebral oxygenation and postoperative cognition recovery for patients undergoing thoracic surgery.

DETAILED DESCRIPTION:
Postoperative neurocognitive impairment is not uncommon for patients undergoing thoracic surgery. Based on the literature, this is associated with reduced cerebral oxygenation during one-lung ventilation which may be because of reduced cardiac output, impeded cerebral venous return due to mechanical ventilation. In our hospital, nonintubated thoracoscopic surgery is commonly conducted and achieves noninferior outcomes than intubated thoracoscopic surgery. Particularly, the application of nasal high flow oxygen may maintain intraoperative oxygenation despite the absence of controlled ventilation. Therefore, the nonintubated technique may be beneficial to maintain an improved intraoperative cerebral oxygenation and hopefully improves postoperative cognition recovery. In this randomized controlled study, we aim to investigate the differences in intraoperative cerebral oxygenation and postoperative cognitive recovery bewteen nonintubated and intubated thoracoscopic surgery. Patient will be randomly assigned to receive nonintubated or intubated thoracoscopic surgery. During surgery, bifrontal cerebral oxygenation will be monitored. Cognitive test will be arranged before and after surgery.

ELIGIBILITY:
Inclusion criteria:

Adult patients receive elective thoracoscopic surgery

Exclusion criteria:

1. pregnancy
2. preexisting cerebral dysfunction such as cerebral vascular incidence, Alzheimer's Disease. Parkinsonism.
3. Cardiopulmonary dysfunction such as heart failure > New York Heart Association score III; chronic obstructive pulmonary disease with a forced expiratory volume in one second/forced vital capacity < 70 % and FEV1 < 50% predicted.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive recovery | 6 months
  Postoperative cognitive recovery assessed by using the Taiwanese quick mild cogntive impairment (Qmci-TW) test (score 0-100) at the baseline (the day before surgery), 24 hour and 6 months after surgery

SECONDARY OUTCOMES:
Intraoperative cerebral oxygenation | throughout surgery; approximately 2.5 hours
  Intraoperative cerebral oxygenation changes during one-lung ventilation will be noninvasively monitored by using near infrared spectroscopy.
Comprehensive complication index | The hospital stayl approximately 3 days
  The comprehensive complication index was calculated in each patient during the hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan